CLINICAL TRIAL: NCT06946095
Title: Efficacy and Safety of Xinyue Capsule in the Treatment of Heart Failure With Preserved Ejection Fraction: A Clinical Study
Brief Title: Efficacy and Safety of Xinyue Capsule in the Treatment of Heart Failure With Preserved Ejection Fraction
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: drjihuang
Record Dates: First submitted 2025-04-09; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Heart Failure
Keywords: Heart Failure with Preserved Ejection Fraction
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chinese patent medicine (Experimental): Add Xinyue Capsules to the regular western medicine treatment.
  Interventions: Drug: Chinese patent medicine
- western medicine treatment (No Intervention): only use the regular western medicine treatment

INTERVENTIONS:
Drug: Chinese patent medicine — This study aims to investigate whether the addition of Xinyue Capsule to conventional Western medical therapy significantly improves cardiac function and reduces the level of heart failure biomarker NT-proBNP in patients with Heart Failure with Preserved Ejection Fraction (HFpEF).
  Arms: Chinese patent medicine

SUMMARY:
The purpose of this study is to evaluate the effect of Xinyue Capsule in the improvement cardiac function and reduction the level of heart failure biomarker NT-proBNP in patients suffering from HF with an ejection fraction greater than or equal to 50%. Researchers will also collect information on how much the heart disease has impact on patient's lives, and how well Xinyue Capsule treatment is tolerated. The study plans to enroll 246 male and female patients of the age of 18 years and above suffering from heart failure with ejection fraction greater than or equal to 50%. Participants will take the study product as oral tablet with a dose 0.6 g Tid daily. Study duration will be up to 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, and signed informed consent provided;
2. Presence of symptoms such as dyspnea (including exertional dyspnea, paroxysmal nocturnal dyspnea, orthopnea), fatigue, poor appetite, and bilateral lower limb edema;
3. Left Ventricular Ejection Fraction (LVEF) ≥ 50%, and meeting at least one of the following criteria:

   * NT-proBNP ≥ 125 ng/L (sinus rhythm) or NT-proBNP ≥ 365 ng/L (atrial fibrillation);

Exclusion Criteria:

1. Usage of Xinyue Capsule or other Chinese patent medicines/herbal remedies aimed at alleviating heart failure symptoms or biomarkers within the past 90 days;
2. Known intolerance or significant allergic reaction to Xinyue Capsule;
3. Occurrence of cardiovascular adverse events within the past 90 days;
4. Acute decompensated heart failure, life-threatening arrhythmias, acute myocardial infarction, or cardiogenic shock;
5. Heart failure secondary to pulmonary hypertension, anemia, thyroid disorders, chronic obstructive pulmonary disease, or musculoskeletal disorders;
6. Presence of cardiac amyloidosis, storage diseases (hemochromatosis, glycogen storage disease), severe valvular heart disease, severe infections, malignancies, or significant hepatic or renal insufficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Estimated)
Dates: Start 2025-05-20 (Estimated); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
N-terminal pro-brain natriuretic peptide (NT-proBNP). | At baseline, Weeks 12

SECONDARY OUTCOMES:
Mitral Annular e' Velocity Mitral Annular e' Velocity: Mitral Annular e' Velocity: | At baseline, Weeks 12
  The mitral annular e' velocity is measured using tissue Doppler imaging (TDI) at the lateral or septal side of the mitral annulus during early diastole. It reflects the relaxation capacity of the left ventricle (LV). Reduced e' velocity is a key indicator of impaired LV diastolic function.
Six-minute walk distance. | At baseline, Weeks 12
  A simple, non-invasive clinical test used to evaluate cardiopulmonary function and exercise tolerance. The patient walks as far as possible on a flat, hard surface for 6 minutes, with the total distance recorded. Longer 6MWD correlates with higher survival rates and lower hospitalization risks, especially in chronic heart or lung disease patients.
Minnesota Living with Heart Failure Questionnaire | At baseline, Weeks 12
  The Minnesota Living with Heart Failure Questionnaire (MLHFQ) is a validated, patient-reported outcome measure specifically designed to assess the impact of heart failure on a patient's quality of life. It consists of 21 items that evaluate physical, emotional, and social limitations caused by heart failure over the preceding 4 weeks.
  The Minnesota Living with Heart Failure Questionnaire (MLHFQ) is a validated, patient-reported outcome measure specifically designed to assess the impact of heart failure on a patient's quality of life. It consists of 21 items that evaluate physical, emotional, and social limitations caused by heart failure over the preceding 4 weeks.
  The Minnesota Living with Heart Failure Questionnaire (MLHFQ) is a validated, patient-reported outcome measure specifically designed to assess the impact of heart failure on a patient's quality of life. The total score ranges from 0 to 105, with higher scores indicating poorer quality of life.
PHQ-9 score | At baseline, Weeks 12
  The Patient Health Questionnaire-9 (PHQ-9) is a widely used screening tool for assessing the presence and severity of depressive symptoms. It consists of 9 questions, each corresponding to a symptom of major depressive disorder as defined by the DSM-5. Scores ≥10 typically indicate clinically significant depression requiring further evaluation. High scores (≥15) or suicidal ideation necessitate urgent referral to mental health professionals.
Average E/e' Ratio | At baseline, Weeks 12
  The E/e' ratio is calculated by dividing the peak early diastolic mitral inflow velocity (E-wave, measured by pulsed-wave Doppler) by the average of the septal and lateral mitral annular e' velocities (from TDI). This ratio is used to estimate left ventricular filling pressure. An elevated E/e' ratio (typically >14) suggests increased diastolic filling pressure and possible heart failure with preserved ejection fraction (HFpEF).
Left Atrial Volume Index (LAVI) | At baseline, Weeks 12
  The left atrial volume index is a measurement of left atrial size, calculated by dividing the left atrial volume (measured via the biplane method of disks on echocardiography) by the patient's body surface area (BSA). Elevated LAVI (>34 mL/m²) indicates left atrial enlargement, which is associated with chronic diastolic dysfunction, atrial fibrillation, and adverse cardiovascular outcomes.
Tricuspid Regurgitation Peak Velocity (TR Vmax) | At baseline, Weeks 12
  The peak velocity of the tricuspid regurgitation jet is measured using continuous-wave Doppler. It reflects the pressure gradient between the right ventricle and right atrium during systole. Elevated TR Vmax (>3.4 m/s) is used to estimate pulmonary artery systolic pressure (using the simplified Bernoulli equation: 4V²) and may indicate pulmonary hypertension.
Left Ventricular Eccentricity Index (LVEI) | At baseline, Weeks 12
  The left ventricular eccentricity index assesses the geometric shape of the LV in short-axis view at end-diastole. It is calculated as the ratio of the anteroposterior diameter to the septolateral diameter of the LV. An index >1.0 indicates LV eccentric remodeling, often seen in volume overload states (e.g., mitral/aortic regurgitation) or adaptive changes in dilated cardiomyopathy. In pressure overload (e.g., aortic stenosis), concentric remodeling typically predominates.
GAD-7 scores | At baseline, Weeks 12
  The Generalized Anxiety Disorder-7 (GAD-7) is a validated screening tool used to assess the presence and severity of generalized anxiety symptoms. It contains 7 questions that align with DSM-5 criteria for generalized anxiety disorder (GAD). Scores ≥10: Refer for further evaluation (e.g., psychological assessment, diagnosis). Scores ≥15 or suicidal thoughts: Prioritize urgent mental health intervention. Monitor patients with chronic conditions (e.g., chronic pain, cancer) who may experience overlapping anxiety symptoms.

IPD SHARING:
Plan to Share IPD: No